CLINICAL TRIAL: NCT03595436
Title: The Effects of Protein Source on Appetite Control, Satiety, and Subsequent Food Intake: A Clinical Screening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1711019935
Record Dates: First submitted 2018-06-30; First posted 2018-07-23 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: tightly-controlled, randomized crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pea Protein Breakfast Preload (Experimental): The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preloads will be standardized to ~325 kcal. The preloads will include the same fat content but will vary in protein and carbohydrate amounts. All ingredients are GRAS listed and approved.
  Interventions: Dietary Supplement: Pea Protein-20g; Dietary Supplement: Pea Protein-30g; Dietary Supplement: Pea Protein-40g
- Carbohydrate Control Breakfast Preload (Placebo Comparator): The study participants will be provided with a control breakfast preload to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. The preload will include the same fat content (as the Experimental Preloads) but will vary in protein and carbohydrate amounts. All ingredients are GRAS listed and approved.
  Interventions: Dietary Supplement: Carbohydrate Control
- Whey Protein (Active Comparator): The study participants will be provided with an active control breakfast preload to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. The preload will include the same fat content (as the Experimental Preloads) but will vary in protein amount and type and carbohydrate amount. All ingredients are GRAS listed and approved.
  Interventions: Dietary Supplement: Whey Protein-20g

INTERVENTIONS:
Dietary Supplement: Pea Protein-20g — The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. This preload will include 20 g pea protein, 5 g mixed protein (from yogurt and peanut-butter), 40 g carbohydrates, and 7 g fat. The preload is a yogurt-based (chocolate-peanut butter flavored) breakfast.
  Arms: Pea Protein Breakfast Preload
Dietary Supplement: Pea Protein-30g — The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. This preload will include 30 g pea protein, 5 g mixed protein (from yogurt and peanut-butter), 32 g carbohydrates, and 7 g fat. The preload is a yogurt-based (chocolate-peanut butter flavored) breakfast.
  Arms: Pea Protein Breakfast Preload
Dietary Supplement: Pea Protein-40g — The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. This preload will include 40 g pea protein, 5 g mixed protein (from yogurt and peanut-butter), 24 g carbohydrates, and 7 g fat. The preload is a yogurt-based (chocolate-peanut butter flavored) breakfast.
  Arms: Pea Protein Breakfast Preload
Dietary Supplement: Whey Protein-20g — The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. This preload will include 20 g whey protein, 5 g mixed protein (from yogurt and peanut-butter), 40 g carbohydrates, and 7 g fat. The preload is a yogurt-based (chocolate-peanut butter flavored) breakfast.
  Arms: Whey Protein
Dietary Supplement: Carbohydrate Control — The study participants will be provided with breakfast preloads to consume. The energy content of the breakfast preload will be standardized to ~325 kcal. This preload will include 5 g mixed protein (from yogurt and peanut-butter), 59 g carbohydrates, and 7 g fat. The preload is a yogurt-based (chocolate-peanut butter flavored) breakfast.
  Arms: Carbohydrate Control Breakfast Preload

SUMMARY:
Primary Objective: To examine whether the consumption of preloads varying in protein quality effect subsequent meal energy and macronutrient content

Secondary Objectives: To examine whether the consumption of preloads varying in protein quality effect postprandial feelings of hunger, fullness, desire to eat, prospective food consumption, and eating initiation.

Exploratory Objective: To examine whether the consumption of preloads varying in protein quality effect postprandial cognitive performance.

DETAILED DESCRIPTION:
The investigators propose the following acute, randomized crossover study to compare 5, isocaloric yogurt-based preloads containing 20, 30, or 40 g pea protein; 20 g whey protein; and an isocaloric carbohydrate (control).

For 3 consecutive days/pattern, the participants will consume the respective treatment, at home, between 7-9 am, based on their habitual breakfast time. (These days are implemented to allow for the acclimation to the respective preload. Using this approach, the participant becomes familiar with the taste profile along with the practice of consuming a breakfast 'shake' so that the testing day more closely assimilates the habitual effects of the preload on appetite, satiety, and food intake.)

On day 4, the participants will report to the research facility 1 h prior to their habitual breakfast time to complete each 4-h testing day. Upon arrival to the facility, each participant will become familiarized with the testing day procedures. At time -15 min, a baseline set of computerized appetite/satiety and cognitive function questionnaires will be completed. At time 0 min, the respective preload will be provided. Immediately following the first swallow of the preload, the participants will be given a questionnaire assessing the palatability. The participants will consume the preload within 10 min. Afterwards, the participants will continue to complete the questionnaires every 30 min throughout the 4-h postprandial period. In addition to these questionnaires, participants will complete a cognitive function paradigm at -30 min, +90 min, and +180 minutes in order to assess memory, executive function, attention, and reaction time. Throughout the day, the participants will also indicate if/when they would like to eat again. Regardless of their meal timing request, at 4-h post-breakfast, lunch will be provided. The participants will be given 30 min to "consume as much or as little as they wish until comfortably full." Following these procedures, the participants will be allowed to leave the facility. There will be a 3-7 day washout period between testing days.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI: 18.0-24.5 kg/m2)
* No history of smoking
* No metabolic or hormonal conditions/diseases that influence metabolism, appetite, or food intake
* No past history of surgical interventions for the treatment of obesity
* No weight loss/gain (≥10 lb. in the past 6 months)
* No medication that would influence directly appetite or cognition
* No change in any medications (over the past 3 months)
* Not currently/previously on a special diet such as Atkins/Ketogenic, high protein, vegan, vegetarian, etc.
* Habitually consumes breakfast (i.e., of at least 350 kcal on ≥ 5 days/wk prior to 9 am
* Habitually consumes lunch (i.e., of at least 350 kcal on ≥ 5 days/wk approximately 4 h after breakfast
* Not clinically diagnosed with an eating disorder such as anorexia, bulimia, night-eating syndrome
* Displays a score of <4 on the Three Factor Eating Habits Questionnaire (TFEQ)
* No allergies and/or aversions to the food/ingredients included within the study
* No history of drug or alcohol abuse (i.e., >14 drinks/week)
* Willing to maintain current activity dietary patterns throughout the study
* Willing to consume all study breakfast and lunch foods
* Generally healthy, as assessed from the medical history questionnaire
* Rating of ≥ 5 illustrating a minimum of "neither like nor dislike on a hedonic 9 pt taste test of the breakfast preloads

Exclusion Criteria:

* Clinically diagnosed with an eating disorder
* Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
* Currently or previously on a weight loss or other special diet (in the past 6 months)
* Gained/lost >10 lb. over the past 6 months
* Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months)
* Not willing or able to complete all study testing procedures

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Perceived Hunger | -30 min, 0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min
  A questionnaire assessing perceived hunger will be completed at specific times throughout each of the the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min hunger) and 100 is max (hunger). A summation (area under the curve) will be calculated.
Perceived Fullness | -30 min, 0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min
  A questionnaire assessing perceived fullness will be completed at specific times throughout each of the the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated.
Perceived Desire to Eat | -30 min, 0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min
  A questionnaire assessing perceived desire to eat will be completed at specific times throughout each of the the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated.
Perceived Prospective Food Consumption | -30 min, 0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min
  A questionnaire assessing how much could be consumed will be completed at specific times throughout each of the the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated.
Lunch Energy Intake | 5 testing days across ~ 2 months
  The participants will be provided with an ad libitum pizza lunch to consume ad libitum. The amount of pizza provided (in grams) will be weight prior to consumption and any remains will be re-weighted after consumption. Energy consumed will be calculated.

SECONDARY OUTCOMES:
Perceived Breakfast Preload Palatability | 5 testing days across ~ 2 months
  A questionnaire assessing how much the breakfast is liked will be completed after the breakfast is meal is started for each of the the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Leidy, PhD, Principal Investigator — Associate Professor
Locations (1):
- Purdue University, West Lafayette, Indiana, United States